CLINICAL TRIAL: NCT01972035
Title: ValGanciclovir Versus ValAcyclovir for Viral Prophylaxis in Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 130162
Record Dates: First submitted 2013-10-10; First posted 2013-10-30 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Transplantation Infection; Epstein-Barr Virus Infections; Cytomegalovirus Infections
Keywords: EBV; CMV; Kidney transplant; valganciclovir; valacyclovir
MeSH Terms: conditions — Epstein-Barr Virus Infections; Cytomegalovirus Infections | interventions — Valacyclovir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ValAcyclovir (Experimental): Kidney recipients who give informed consent will be randomly assigned to receive ValA or ValG in a 1:1 ratio. Duration of therapy is 3-12 months depending on risk and age of recipient. Dosing is based on glomerular filtration rate.
  Interventions: Drug: Valacyclovir
- ValGanciclovir (Active Comparator): Kidney recipients who give informed consent will be randomly assigned to receive ValG or ValA in a 1:1 ratio. Duration of therapy is 3-12 months depending on risk and age of recipient. Dosing is based on glomerular filtration rate.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valacyclovir — Experimental Arm
  Other Names: Valtrex; Valacyclovir Hydrochloride; Valacyclovir HCL
  Arms: ValAcyclovir
Drug: Valganciclovir — Standard of care
  Other Names: Valcyte; Valganciclovir hydrochloride
  Arms: ValGanciclovir

SUMMARY:
Our study will compare all kidney transplant recipients receiving valganciclovir vs. valacyclovir for one year following kidney transplant and compare:

1. the incidence, magnitude and duration of CMV and EBV viremia in the first year after transplant.
2. the side effects of the anti-viral drugs requiring dose reduction or cessation

In addition, we will test renal tissue obtained from any biopsies post-transplant (surveillance or clinically indicated biopsies) by both polymerase chain reaction (PCR) and fluorescence in situ hybridization to assess for latent CMV and/or EBV.

DETAILED DESCRIPTION:
Herpes viruses such as Epstein-Barr virus (EBV) and cytomegalovirus (CMV) cause considerable morbidity and mortality post-kidney transplant. Even subclinical CMV and/or EBV viremia have been associated with deterioration in kidney transplant function. Currently, valganciclovir (valG) is the primary prophylactic agent against CMV in kidney transplant recipients but CMV viremia has been noted in 22% of pediatric post-kidney transplant recipients, and the incidence at the University of Minnesota (UMMC) in all kidney transplant recipients is as high as 17% despite valG prophylaxis. CMV disease post-kidney transplant can manifest as fever, leucopenia, or mild to severe organ involvement. While an effective anti-CMV drug, valG has a number of adverse effects including leucopenia, also a side effect of mycophenolate mofetil (MMF), one of the cornerstones of current anti-rejection regimens. Combined therapy with MMF and valG frequently results in leucopenia associated infection or leucopenia necessitating reduction in MMF doses, increasing the risk of rejection. In addition, valG is prohibitively expensive forcing many centers adopt a pre-emptive therapeutic approach whereby post-Ktx patients are screened for CMV, and at new onset viremia, valG is initiated. This approach has been associated with increased CMV infections and resistant viral strains. Therefore, there is need for an alternate, more cost-effective drug with a more benign side effect profile and equal effectiveness against CMV.

To date, the anti-EBV effect of valG is poorly defined and prevention of EBV infection is by close monitoring and immunosuppression reduction at the discovery of EBV viremia. EBV can present post-kidney transplants as infectious mononucleosis syndrome, hepatitis and, most importantly, can initiate potentially fatal lymphoproliferative disorders (PTLD). Between October 2003 and December 2009, EBV viremia occurred in 20% of adults and 50% of pediatric kidney transplant recipients (60/120) at UMMC, and, PTLD occurred in 6% (7/120) of pediatric recipients. Effective anti-EBV prophylaxis could substantially improve kidney transplant outcomes.

UMMC conducts surveillance biopsies at transplant and 3 and 12 months post-kidney transplant on all adult transplant recipients, providing an ideal opportunity to assess kidney tissue for EBV and CMV via molecular and immunological assays. Isolating the virus from infected recipient would be a pivotal step in our understanding of the mechanisms of CMV and EBV infection post-kidney transplant.

In summary, if valacyclovir and valganciclovir have equivalent efficacy in CMV prophylaxis, and valacyclovir has the anticipated effect on EBV prevention, the use of valacyclovir will result in a reduced risk of leucopenia-associated infection, and a lower incidence of rejection by allowing the use of standard MMF doses. Since valacyclovir is cheaper, it is plausible that universal prophylaxis will be a plausible and affordable option for all transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* All consenting kidney transplant recipients.

Exclusion Criteria:

* Non-consent.
* Recipients with allergies to valacyclovir or valganciclovir
* Recipients that are unable to independently understand the consent form and do not have a legally authorized representative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hank Balfour, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Kacer M, Kielberger L, Bouda M, Reischig T. Valganciclovir versus valacyclovir prophylaxis for prevention of cytomegalovirus: an economic perspective. Transpl Infect Dis. 2015 Jun;17(3):334-41. doi: 10.1111/tid.12383. Epub 2015 May 26. PMID 25824586
- [Background] Reischig T, Kacer M, Jindra P, Hes O, Lysak D, Bouda M. Randomized trial of valganciclovir versus valacyclovir prophylaxis for prevention of cytomegalovirus in renal transplantation. Clin J Am Soc Nephrol. 2015 Feb 6;10(2):294-304. doi: 10.2215/CJN.07020714. Epub 2014 Nov 25. PMID 25424991

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ValAcyclovir | ValGanciclovir
Started | 66 | 71
Completed | 27 | 44
Not Completed | 39 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ValAcyclovir | ValGanciclovir | Total
Number analyzed (Participants) | 66 | 71 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 19 | 41
  Between 18 and 65 years | 44 | 52 | 96
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 40 | 42 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 53 | 58 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 66 | 71 | 137

OUTCOME MEASURES:

1. Primary Outcome: Compare Incidence, Duration and Magnitude of CMV and EBV Viremia in Kidney Transplant Recipients Receiving valA vs. valG.
Description: In infectious mononucleosis intervention trials, two weeks of valA therapy resulted in a statistically significant reduction in oral EBV shedding, accompanied by a clinical benefit, and valA is currently used for the therapy of severe cases of infectious mononucleosis in the community. ValA has also been shown to reduce the incidence and delay the onset of CMV disease in both CMV seronegative patients (P<0.001) and CMV seropositive patients (P=0.03). Therefore we hypothesize that the anti-EBV and anti-CMV effects of valA will be equal to or more effective than valG in reducing post-kidney transplant EBV and CMV viremia.
Time Frame: First year post-kidney transplant
Measure: Count of Participants; unit: Participants
Arm/Group | ValAcyclovir | ValGanciclovir
Number analyzed (Participants) | 66 | 71
Participants
  EBV Viremia | 16 | 20
  CMV Viremia | 8 | 4
  BK Viremia | 5 | 11
  PTLD/EBV Disease | 2 | 1
  None | 35 | 35

ADVERSE EVENTS:
Time Frame: 1 year following intervention
Arm/Group | ValAcyclovir | ValGanciclovir
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/71
Serious Adverse Events (participants affected / at risk) | 52/66 | 50/71
Other Adverse Events (participants affected / at risk) | 64/66 | 70/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ValAcyclovir (N=66) | ValGanciclovir (N=71)
Acute Kidney Problems (Renal and urinary disorders) | 3 (3) | 3 (3)
Ascites (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Bacterial Infection (Infections and infestations) | 1 (1) | 2 (2)
Biopsy (Investigations) | 5 (5) | 3 (3)
Blood sugar concerns (Endocrine disorders) | 1 (1) | 2 (2)
Breathing concerns (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Donor source antibodies (Immune system disorders) | 4 (4) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 21 (21) | 21 (23)
Fever (Immune system disorders) | 7 (9) | 7 (9)
G Tube Concerns (Surgical and medical procedures) | 1 (3) | 3 (9)
Heart concerns (Cardiac disorders) | 6 (7) | 5 (5)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Mental Concerns (Psychiatric disorders) | 0 (0) | 2 (4)
Severe Pain (General disorders) | 9 (11) | 4 (4)
Thrombosis (Vascular disorders) | 3 (3) | 4 (4)
Upper Respiratory Infection (Immune system disorders) | 7 (9) | 6 (10)
Urination Concerns (Renal and urinary disorders) | 3 (4) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 6 (10) | 11 (19)
Other (General disorders) | 10 (12) | 10 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ValAcyclovir (N=66) | ValGanciclovir (N=71)
Abdominal Pain (Gastrointestinal disorders) | 21 | 20
Diarrhea (Gastrointestinal disorders) | 43 | 46
Nausea (Gastrointestinal disorders) | 25 | 28
Emesis (Gastrointestinal disorders) | 23 | 31
Fatigue (General disorders) | 8 | 8/11
Alopecia (Immune system disorders) | 1 | 3
Anemia (Blood and lymphatic system disorders) | 64 | 70
Abnormal LFTs (Hepatobiliary disorders) | 2 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 46
Headache (General disorders) | 6 | 11
Peripheral neuropathy (Nervous system disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT01972035/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT01972035/ICF_000.pdf